CLINICAL TRIAL: NCT06984965
Title: Role of Electroencephalogram (EEG) in Differentiation Between Ischemic and Hemorrhagic Stroke and as a Predictor of Post-stroke Recovery
Brief Title: Role of EEG in Differentiation Between Ischemic and Hemorrhagic Stroke
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gena ELassall, Residant at Neurology Department, Faculty of Medicine, Assiut University, Assiut University
Other Study IDs: 04-2024-200998
Record Dates: First submitted 2024-12-28; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-01

CONDITIONS: Acute Ischemic Stroke; Acute Haemorrhagic Stroke
Keywords: EEG; Acute Ischaemic Stroke; Acute Haemorrhagic Stroke; Stroke Recovery
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Ischaemic Stroke Group: Patients with ischemic arteria cerebri media infarct confirmed by MRI.
- Haemorrhagic Stroke Group: Patients with spontaneous intraparenchymal bleeding confirmed by CT.

SUMMARY:
Searching electrical activity registered by EEG in acute ischemic and hemorrhagic stroke and comparing these parameters to the poststroke recovery patterns to investigate the role of EEG as a differentiation tool and as a predictor of post-stroke recovery.

DETAILED DESCRIPTION:
In this study, EEG will be performed on each patient included; within 72 hours of the onset of the stroke. The EEG device will be used within the intended use as described in the user manuals. The electrodes are put on the patient's head, and the EEG signal is recorded for several minutes; the amplifier is used to amplify the EEG signal and reduce artifacts. A complete EEG and data will be collected at baseline and on follow-up to observe the differences in EEG patterns to perform a qualitative assessment of the EEG results.

EEG patterns depend on the size and location of acute ischemic stroke, including generalized or focal slowing or both and epileptiform discharges. Abnormal neuronal activity is determined by comparing a part of the patient's brain not affected by stroke to a part of the patient's brain affected by stroke. Moreover, Abnormal blood flow is interpreted by comparing the abnormal EEG patterns in the areas of infarctions or hemorrhage to the normal brain tissue signals. The aim is to compare electric waveforms from an EEG device between patients with acute ischemic and acute hemorrhagic stroke (at baseline which is within 72 hours of the onset of acute ischemic and acute hemorrhagic stroke and through study completion, an average of 3 to 6 months).

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 and below 80 years.
* Acute Ischemic stroke: ischemic arteria cerebri media infarct confirmed by MRI.
* Acute Hemorrhagic stroke: spontaneous intraparenchymal bleeding confirmed by CT.
* Stroke onset <72 hours before expected time of performing EEG.
* First-ever ischemic stroke.
* Measurable deficit on the National Institute of Health Stroke Scale (NIHSS).
* Able to give and sign informed consent.

Exclusion Criteria:

* Transient Ischemic Attacks (TIAs).
* Greater than 72 hours past the initial insult.
* Patients with subarachnoid haemorrhage, traumatic haemorrhage (epidural/subdural bleeding), cerebral venous sinus thrombosis, indication for urgent neurosurgical intervention.
* History of other central nervous system diseases.
* Any signs unfit for MRI/EEG scan.
* Injury or active infection of electrode cap placement area.
* Claustrophobia; recognition disorder.
* Known skull defect or head trauma.
* Previous neurological procedure (metallic implant, brain pace, cranial operation history).
* Significant physical impairment that would restrict the ability to use the portable EEG devices.
* Presence of malignancy or systemic rheumatic disease
* Non-stroke disease or lesion affecting the sensorimotor system.
* Alcohol or drug addiction.
* Presence of pump/shunt.
* Presence of Malignancy.
* Presence of severe cognitive impairment.
* History of epilepsy or taking medication due to epilepsy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute Ischemic stroke: ischemic arteria cerebri media infarct confirmed by MRI, or acute Hemorrhagic stroke: spontaneous intraparenchymal bleeding confirmed by CT, onset <72 hours before expected time of performing EEG.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants With Focal Slowing in the Stroke-Affected Hemisphere | Baseline (within 72 hours of stroke onset)
  Presence of focal slowing (e.g., increased delta or theta activity) in the stroke-affected hemisphere versus the unaffected hemisphere. Patterns categorized as "ischemic" or "hemorrhagic."; this will be measured in percentage (%).
Proportion of Participants With Interhemispheric Asymmetry in EEG Waveforms | Baseline (within 72 hours of stroke onset)
  Qualitative assessment of EEG asymmetry between affected and unaffected hemispheres at baseline. Frequency of each will be measured in percentage (%).
Proportion of Participants With Absent or Diminished EEG Reactivity | Baseline (within 72 hours of stroke onset)
  Absence or reduction in EEG reactivity to external stimuli (e.g., auditory, tactile) in the affected hemisphere; this will be measures by precentage (%).
Proportion of Participants With Epileptiform Activity on EEG | Baseline (within 72 hours of stroke onset)
  Presence of epileptiform discharges (e.g., spikes or sharp waves) on EEG in the stroke-affected hemisphere; thsi will be measured by precentage (%).

SECONDARY OUTCOMES:
Correlation Between Baseline EEG Findings and Functional Recovery | Phase I (Baseline EEG assessment) and Phase III (3 to 6 month follow-up functional evaluation)
  Association between initial qualitative EEG abnormalities (e.g., focal slowing, asymmetry) and functional outcomes measured by standardized scales (e.g., Modified Rankin Scale) at 6 months; measured by Correlation coefficient (r).
Prediction of Post-Stroke Seizures Based on EEG Findings | Phase I (Baseline EEG assessment) and Phase III (3 to 6 month follow-up functional evaluation)
  Proportion of participants with specific EEG abnormalities (e.g., epileptiform activity) at baseline who develop post-stroke seizures within 3 to 6 months, measured by percentage (%).

CONTACTS AND LOCATIONS:
Locations (1):
- Neurology Department, Faculty of Medicine, Assiut University, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided